CLINICAL TRIAL: NCT00959582
Title: A Multicenter Trial to Measure Early Patterns of Change in [18F]-Fluorodeoxyglucose Uptake by PET/CT in Relapsed Ovarian Cancer Patients
Brief Title: Positron Emission Tomography/Computed Tomography (PET/CT) in Relapsed Ovarian Cancer (MK-0000-143)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0000-143; 2009_632
Record Dates: First submitted 2009-08-12; First posted 2009-08-14 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Relapsed ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 18-F-FDG PET/CT imaging
  Interventions: Procedure: Comparator: 18-F-FDG PET/CT and Volumetric CT

INTERVENTIONS:
Procedure: Comparator: 18-F-FDG PET/CT and Volumetric CT — Patients will receive standard-of-care therapy (carboplatin or cisplatin monotherapy, or a two-drug combination where one is platinum). FDG-PET/CT scans will be performed at baseline following enrollment, after Cycles 1 and 2 of chemotherapy, and if patients are progression-free at the end of Cycle 6. Volumetric CT scans will be performed at baseline following enrollment, after Cycles 1 and 2 of chemotherapy, after Cycle 3 of chemotherapy (optional), and if patients are progression-free at the end of Cycle 6 and at 40 weeks after Cycle 1 dosing.

SUMMARY:
This study will characterize FDG-PET (18F-Fluorodeoxyglucose-Positron Emission Tomography) as an early response marker in recurrent, platinum-sensitive ovarian cancer treated with platinum-based therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient has ovarian, primary peritoneal, or fallopian tube cancer
* Patient has first or subsequent relapse
* Patient has had at least on prior platinum-based treatment for ovarian cancer
* Patient is scheduled to receive treatment with carboplatin or cisplatin monotherapy or combination where one of the drugs is a platinum
* Patient is not pregnant

Exclusion Criteria:

* Patient has had abdominal surgery within the last 6 weeks
* Patient has life expectancy < 6 months
* Patient has had radiotherapy to the abdomen or pelvis within the last 6 months
* Patient has poorly controlled diabetes

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with metabolic non-response assessed by FDG-PET standardized uptake value (SUV) 3 weeks and 6 weeks after starting platinum-based therapy | Baseline, Week 3, Week 6
Progression free proportion | 40 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC